CLINICAL TRIAL: NCT00429208
Title: Effect Of Nicotine on Neurocognitive Performance of Cigarette Smokers: A Double-Blind, Within-Subjects, Placebo-Controlled Study
Brief Title: Effect Of Nicotine on Neurocognitive Performance of Cigarette Smokers
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hadassah Medical Organization (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: Double | Purpose: Diagnostic
Other Study IDs: yakir@hmo
Record Dates: First submitted 2007-01-30; First posted 2007-01-31 (Estimated); Last update posted 2007-01-31 (Estimated); Status verified 2007-01

CONDITIONS: Nicotine Dependence; Smoking; Tobacco Use Disorder; Nicotine Use Disorder
Keywords: Nicotine Dependence; Smoking; Tobacco Use Disorder; Nicotine Use Disorder
MeSH Terms: conditions — Tobacco Use Disorder; Smoking | interventions — Nicotine

INTERVENTIONS:
Drug: Nicotine

SUMMARY:
This research project addresses the hypothesis that a neurocognitive profile characterized by impairment of response inhibition and sustained attention may be a risk factor for smoking initiation and nicotine dependence among young women. Nicotine has short- term, facilitating effects on attention and response inhibition. Therefore, individuals who are impaired on cognitive functions such as these and initiate cigarette smoking may be more likely to maintain the habit and develop nicotine dependence. The research protocol specifically tests whether administration of nicotine to non-abstinent, regular cigarette smokers improves cognitive function in those domains where the participants had previously been shown to manifest performance deficits

ELIGIBILITY:
Inclusion Criteria:

* Reported smoking cigarettes on a daily basis at the time of the original study and continue to smoke currently
* Manifested poor performance on the MFFT (The neurocognitive test that yielded differences between smokers and non-smokers)
* Competent and willing to give written informed consent

Exclusion Criteria:

* Pregnancy, breast-feeding, non-use of contraception such that the possibility of pregnancy cannot be excluded
* Intake of any medication that may potentially interact with nicotine.
* Any current or past medical condition that represents a contra-indication to nicotine administration.

Ages: 18 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2007-02; Study Completion 2007-04 (Estimated)

PRIMARY OUTCOMES:
Neurocognitive functions

CONTACTS AND LOCATIONS:
Overall Officials: Avi Yakir, MD, Principal Investigator — Hadassah Medical Organization
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel

REFERENCES:
- [Result] Yakir A, Rigbi A, Kanyas K, Pollak Y, Kahana G, Karni O, Eitan R, Kertzman S, Lerer B. Why do young women smoke? III. Attention and impulsivity as neurocognitive predisposing factors. Eur Neuropsychopharmacol. 2007 Apr;17(5):339-51. doi: 10.1016/j.euroneuro.2006.09.004. Epub 2006 Nov 30. PMID 17141485